CLINICAL TRIAL: NCT05492981
Title: Does an Educational Video for Aneuploidy Screening Improve Informed Choice Among Pregnant Women? A Randomized Controlled Trial
Brief Title: Does an Educational Video for Aneuploidy Screening Improve Informed Choice Among Pregnant Women?
Acronym: EVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020/01123
Record Dates: First submitted 2022-07-31; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Aneuploidy; Down Syndrome; Pregnancy Early
Keywords: prenatal; Screening; informed choice; randomized controlled trial
MeSH Terms: conditions — Aneuploidy; Down Syndrome | interventions — Methods; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention was a 16-minute educational video created by the study investigators which provided information about Down syndrome, diagnostic tests and screening tests. The screening tests covered in the video included the triple test, the combined first trimester screen and non-invasive prenatal screening. Information about how and when each of the tests were performed, their detection rates and possible results and their interpretations were covered in the video. The video was viewed by several healthcare providers and experts in the field of prenatal screening before the commencement of this study to ensure that the content was appropriate and adequate. The intervention was viewed by subjects on a portable tablet in a quiet room in the antenatal clinic. Subjects were then invited to ask their doctor any questions that they may have had about the video during the clinic consult which followed.
  Interventions: Behavioral: Enhanced (intervention) education
- Control (No Intervention): Women in the control group were counselled by the referring doctor regarding the aneuploidy screening options of FTS or NIPS, and provided information about the procedures involved for each test, their detection rates, cost, and possible results of testing. The use of a written information leaflet was available to doctors as an adjunct to providing this information.

INTERVENTIONS:
Behavioral: Enhanced (intervention) education — See arm description
  Arms: Intervention

SUMMARY:
Informed decision-making regarding aneuploidy screening has been reported to be low. Poor knowledge and the lack of deliberation have been cited as reasons for uninformed choices, highlighting the need for adequate pre-test counselling. We conducted a study to assess if an educational video improves informed choice in a clinical setting where both the combined first trimester screen and non-invasive prenatal screening are offered routinely to pregnant women.

DETAILED DESCRIPTION:
Women attending the antenatal clinic with a viable singleton pregnancy below 14 weeks were randomized to receive routine counselling by their obstetrician or the intervention, where they watched a 16-minute educational video on aneuploidy screening before their consult. The primary outcome, rate of informed choice, was assessed using an adapted multidimensional measure of informed choice (MMIC) questionnaire, where informed choice was defined as good knowledge and value-consistent behaviour. Secondary outcomes included informed choice with deliberation, decisional conflict and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* aged 21 years or older
* English speaking
* had a viable singleton pregnancy below 14 weeks gestation

Exclusion Criteria:

* women who had any prior discussion with a clinician regarding aneuploidy screening for their current pregnancy

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 286 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Informed choice | Day 0
  Outcome will be measured using the modified multidimensional measure of informed choice (MMIC).

SECONDARY OUTCOMES:
Deliberation | Day 0
  Outcome will be measured using 6 questions to measure deliberation on a five-point Likert scale
Knowledge | Day 0
  Outcome will be measured using a 19-item validated true/false knowledge questionnaire.
Value-consistent behaviour | Day 0
  Attitudes towards testing options were assessed using a validated questionnaire and deemed to be value consistent if a participants had a positive attitude towards the test option that they chose, or a negative attitude towards all test options and chose not to test.
anxiety | Day 0
  Anxiety was assessed using the Spielberger State trait anxiety inventory (STAI-6) short form which consisted of 6 items
Decisional Conflict | Day 0
  Decisional conflict was measured using a validated Decisional Conflict Scale (DCS)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xian Lim KM, Lewis C, Wong HC, Chong GSL, Gosavi A, Choolani MA. Does an educational video for aneuploidy screening improve informed choice among pregnant women? A randomised controlled trial. Prenat Diagn. 2023 Jan;43(1):42-50. doi: 10.1002/pd.6279. Epub 2022 Dec 28. PMID 36550063